CLINICAL TRIAL: NCT03042975
Title: Imaging Genetics of Laryngeal Dystonia
Status: Recruiting | Type: Observational
Sponsor: Kristina Simonyan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Kristina Simonyan, Professor of Otolaryngology - Head & Neck Surgery, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Other Study IDs: 2019P001576; R01DC011805 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Dystonia; Unaffected Relatives of Laryngeal Dystonia Patients; Voice Tremor; Muscle Tension Dysphonia
Keywords: dystonia; spasmodic dysphonia; imaging; genetics
MeSH Terms: conditions — Dysphonia; Dystonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Brain images and blood samples will be collected. The DNA will be extracted and banked for genetic studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Laryngeal Dystonia: Patients with laryngeal dystonia will undergo an MRI of the brain and a blood draw.
  Interventions: Other: MRI; Procedure: Blood draw
- Unaffected relatives of laryngeal dystonia patients: Unaffected relatives of patients with laryngeal dystonia will undergo an MRI of the brain and a blood draw.
  Interventions: Other: MRI; Procedure: Blood draw
- Voice tremor: Patients with voice tremor will undergo an MRI of the brain and a blood draw.
  Interventions: Other: MRI; Procedure: Blood draw
- Muscle tension dysphonia: Patients with muscle tension dysphonia will undergo an MRI of the brain and a blood draw.
  Interventions: Other: MRI; Procedure: Blood draw

INTERVENTIONS:
Other: MRI — Functional and structural MRI of the brain will be conducted to identify disorder specific neural markers
Procedure: Blood draw — Blood samples will be collected, the DNA will be extracted and banked for genetic studies.

SUMMARY:
The contribution of genetic risk factors to the development of focal dystonias is evident. However, understanding of how variations in the causative gene expression lead to variations in brain abnormalities in different phenotypes of dystonia (e.g., familial, sporadic) remains limited. The research program of the investigators is set to determine the relationship between brain changes and genetic risk factors in laryngeal dystonia (or spasmodic dysphonia). The researchers use a novel approach of combined imaging genetics, next-generation DNA sequencing, and clinical-behavioral testing. The use of a cross-disciplinary approach as a tool for the discovery of the mediating neural mechanisms that bridge the gap from DNA sequence to the pathophysiology of dystonia holds a promise for the understanding of the mechanistic aspects of brain function affected by risk gene variants, which can be used reliably for the discovery of associated genes and neural integrity markers for this disorder. The expected outcome of this study may lead to better clinical management of this disorder, including its improved detection, accurate diagnosis, and assessment of the risk of developing dystonia in family members.

DETAILED DESCRIPTION:
Laryngeal dystonia (LD), or spasmodic dysphonia, is an isolated focal dystonia characterized by selective impairment of speech production due to involuntary spasms in the laryngeal muscles. Despite the well-characterized clinical features of LD, its clinical management remains challenging due, in part, to the absence of objective measures (biomarkers) for early detection and differential diagnosis. This results in diagnostic inaccuracies, which have a negative impact on the patient's quality of life and healthcare costs. Importantly, delayed diagnosis leads to deferred treatment. The objective of this application is to conduct a series of studies that combine advanced machine-learning with neuroimaging and genetics to (1) identify the neural markers that accurately differentiate LD between its clinical phenotypes (adductor vs. abductor), genotypes (sporadic vs. familial), and comorbid disorders (voice tremor and muscle tension dysphonia); (2) determine the early predictive neural markers of LD development in at-risk individuals, and (3) validate associated LD gene mutations. Supported by our preliminary data, our central hypothesis is that brain abnormalities are shaped, in part, by underlying genetic factors and exhibit LD form-characteristic features, which can be used as differential diagnostic and early predictive biomarkers of this disorder. This research is innovative both conceptually and methodologically because it uses a cross-disciplinary approach to focus on the neural pathophysiology and genetic susceptibility factors for LD diagnostic and predictive biomarker discovery. The proposed research is significant because it will directly contribute to closing the critically existing gap in the clinical management of LD. Identification of LD neural and genetic markers is expected to have a positive translational impact by establishing enhanced criteria for accurate differential diagnosis and screening of persons at risk. In short, the successful completion of these studies will open new horizons for the clinical management of LD patients.

ELIGIBILITY:
Inclusion criteria:

1. Males and females of diverse racial and ethnic background, with age across the lifespan;
2. Laryngeal Dystonia patients

   * phenotype: adductor or abductor
   * genotype: familial or sporadic
3. Voice Tremor patients

   * essential or
   * dystonic
4. Muscle tension dysphonia patients
5. Unaffected relatives of laryngeal dystonia patients with

   * familial laryngeal dystonia
   * early-onset laryngeal dystonia (onset at ≤ 35 y.o.)
   * typical onset laryngeal dystonia (onset at ≥ 40 y.o.)
6. Native English speakers.
7. Right-handedness.
8. Normal cognitive status.

Exclusion criteria:

1. Subjects who are incapable of giving informed consent.
2. Pregnant or breastfeeding women until a time when they are no longer pregnant or breastfeeding.
3. Subjects with past or present medical history of (a) major neurological problems, such as stroke, movement disorders (other than LD and VT in the patient groups), brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence; (b) psychiatric problems, such as schizophrenia, bipolar depression, obsessive-compulsive disorder; (c) laryn¬geal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis.
4. Patients who are not symptomatic due to treatment with botulinum toxin injections into the laryngeal muscles.
5. Subjects who receive medication(s) affecting the central nervous system.
6. Subjects with a history of major brain and/or laryngeal surgery.
7. Subjects who have tattoos, ferromagnetic objects in their bodies that cannot be removed for imaging study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: laryngeal dystonia unaffected relatives of laryngeal dystonia patients voice tremor muscle tension dysphonia
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Brain changes in laryngeal dystonia | 5 years
  Identify imaging biomarker of laryngeal dystonia

SECONDARY OUTCOMES:
Genes responsible for laryngeal dystonia | 5 years
  Identify genetic mutations responsible for laryngeal dystonia

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Battistella G, Termsarasab P, Ramdhani RA, Fuertinger S, Simonyan K. Isolated Focal Dystonia as a Disorder of Large-Scale Functional Networks. Cereb Cortex. 2017 Feb 1;27(2):1203-1215. doi: 10.1093/cercor/bhv313. PMID 26679193
- [Result] Vulinovic F, Schaake S, Domingo A, Kumar KR, Defazio G, Mir P, Simonyan K, Ozelius LJ, Bruggemann N, Chung SJ, Rakovic A, Lohmann K, Klein C. Screening study of TUBB4A in isolated dystonia. Parkinsonism Relat Disord. 2017 Aug;41:118-120. doi: 10.1016/j.parkreldis.2017.06.001. Epub 2017 Jun 10. PMID 28655586
- [Result] Termsarasab P, Ramdhani RA, Battistella G, Rubien-Thomas E, Choy M, Farwell IM, Velickovic M, Blitzer A, Frucht SJ, Reilly RB, Hutchinson M, Ozelius LJ, Simonyan K. Neural correlates of abnormal sensory discrimination in laryngeal dystonia. Neuroimage Clin. 2015 Oct 30;10:18-26. doi: 10.1016/j.nicl.2015.10.016. eCollection 2016. PMID 26693398
- [Result] Fuertinger S, Horwitz B, Simonyan K. The Functional Connectome of Speech Control. PLoS Biol. 2015 Jul 23;13(7):e1002209. doi: 10.1371/journal.pbio.1002209. eCollection 2015 Jul. PMID 26204475
- [Result] Simonyan K, Fuertinger S. Speech networks at rest and in action: interactions between functional brain networks controlling speech production. J Neurophysiol. 2015 Apr 1;113(7):2967-78. doi: 10.1152/jn.00964.2014. Epub 2015 Feb 11. PMID 25673742
- [Result] Battistella G, Fuertinger S, Fleysher L, Ozelius LJ, Simonyan K. Cortical sensorimotor alterations classify clinical phenotype and putative genotype of spasmodic dysphonia. Eur J Neurol. 2016 Oct;23(10):1517-27. doi: 10.1111/ene.13067. Epub 2016 Jun 27. PMID 27346568
- [Result] Putzel GG, Fuchs T, Battistella G, Rubien-Thomas E, Frucht SJ, Blitzer A, Ozelius LJ, Simonyan K. GNAL mutation in isolated laryngeal dystonia. Mov Disord. 2016 May;31(5):750-5. doi: 10.1002/mds.26502. Epub 2016 Feb 1. PMID 27093447
- [Result] Rittiner JE, Caffall ZF, Hernandez-Martinez R, Sanderson SM, Pearson JL, Tsukayama KK, Liu AY, Xiao C, Tracy S, Shipman MK, Hickey P, Johnson J, Scott B, Stacy M, Saunders-Pullman R, Bressman S, Simonyan K, Sharma N, Ozelius LJ, Cirulli ET, Calakos N. Functional Genomic Analyses of Mendelian and Sporadic Disease Identify Impaired eIF2alpha Signaling as a Generalizable Mechanism for Dystonia. Neuron. 2016 Dec 21;92(6):1238-1251. doi: 10.1016/j.neuron.2016.11.012. Epub 2016 Dec 8. PMID 27939583
- [Result] Bianchi S, Battistella G, Huddleston H, Scharf R, Fleysher L, Rumbach AF, Frucht SJ, Blitzer A, Ozelius LJ, Simonyan K. Phenotype- and genotype-specific structural alterations in spasmodic dysphonia. Mov Disord. 2017 Apr;32(4):560-568. doi: 10.1002/mds.26920. Epub 2017 Feb 10. PMID 28186656
- [Result] Fuertinger S, Simonyan K. Connectome-Wide Phenotypical and Genotypical Associations in Focal Dystonia. J Neurosci. 2017 Aug 2;37(31):7438-7449. doi: 10.1523/JNEUROSCI.0384-17.2017. Epub 2017 Jul 3. PMID 28674168
- [Derived] de Lima Xavier L, Simonyan K. The extrinsic risk and its association with neural alterations in spasmodic dysphonia. Parkinsonism Relat Disord. 2019 Aug;65:117-123. doi: 10.1016/j.parkreldis.2019.05.034. Epub 2019 May 24. PMID 31153765